CLINICAL TRIAL: NCT06876389
Title: Effect of Multi Strain Probiotic on Ferritin Levels in Children with Iron Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Zulyudisiawan Muin, Pediatric resident, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UH24040220
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Iron Deficiency (ID)
MeSH Terms: conditions — Iron Deficiencies | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Children with Iron deficiency who receive iron standard therapy and probiotic multi strain 2 capsules per day for 30 days
  Interventions: Dietary Supplement: Probiotic
- Group B (Placebo Comparator): Children with Iron deficiency who receive iron standard therapy and placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — In group A, children with iron deficiency received standard therapy. This group was given standard therapy in the form of elemental Fe 3 mg/kgBB/day/orally and L Bio as 2 packs per day and Saccharomyces boulardii given 2 capsules per day (dose 2 x 250 mg or 2 x (2.5 x109 cells/cfu)) for ages 1 year - 18 years for 30 days.
  Arms: Group A
Other: Placebo — In group B, children with iron deficiency received standard therapy with placebo. This group was given standard therapy in the form of elemental Fe 3 mg/kgBB/day/orally and placebo for 30 days.
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to learn about the effect of multi-strain probiotic (bacteria and yeast) on ferritin levels in children age 1 - 18 years old who had iron deficiency in 15 orphanages of Makassar city. The main questions it aims to answer are:

• Are ferritin levels in iron deficiency children given iron standard therapy with multi-strain probiotics (bacteria and yeast) higher than those given iron standard therapy with placebo? Researchers will compare iron standard therapy with multi-strain probiotics (bacteria and yeast) to a placebo to see if muti-strain probiotics works to treat iron deficiency in children.

Participant will :

* Take iron standard therapy with multi-strain probiotics (bacteria and yeast) or iron standard therapy with placebo every day for 30 days
* Ferritin levels were evaluated on day 31

DETAILED DESCRIPTION:
The aim of this study was to assess the effect of multi-strain probiotic (bacteria and yeast) on ferritin levels in children with iron deficiency treatment. It is a randomized controlled trial (RCT) conducted in 15 orphanages of Makassar city in children aged 1 - 18 years. The study population was children aged 1 - 18 years who had iron deficiency. Eligible children are randomized into two groups - an intervention group receiving standard iron therapy with multi-strain probiotics (bacteria and yeast) and a control group receiving standard therapy with placebo. The primary outcome is serum ferritin levels, measured at baseline and after 30 days of intervention. Blood samples are collected to measure ferritin levels. The study aims to enroll 80 infants (40 per group) to detect a clinically meaningful difference in ferritin levels between groups. This trial will provide evidence on whether multi strain probiotic can increasing ferritin levels in children with iron deficiency treatment. The results may inform clinical practice regarding the use of probiotics multi strain as an adjunctive therapy for iron deficiency in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with iron deficiency
* Age 1 year - 18 years
* The parent or person in charge of the foundation signed the informed consent that the child was willing to be included in the study.

Exclusion Criteria:

* Iron deficiency children with infection, renal impairment and hepatic impairment were identified through interviews with caregivers and physical examination of the children.
* Children with immunocompromise (malignancy, malnutrition, HIV).
* Iron deficiency children who have received iron therapy and last consumed 3 months prior to the study.
* Iron deficiency children who were temporarily receiving iron therapy or iron supplementation.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Ferritin level | Ferritin level was measured after 30th days of intervention
  We compare the ferritin levels between children with iron deficiency who received standard iron therapy with probiotic multi-strain and those who received standard iron therapy with placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided